CLINICAL TRIAL: NCT00140985
Title: A Randomized, Parallel, Double Blind Study of Losartan Versus Amlodipine in Patients With Mild to Moderate Hypertension and Chronic Nondiabetic Proteinuric Nephropathy: Evaluation of the Effect on Proteinuria and on the Plasmatic Levels of Growth Factors (TGFß and VEGF)
Brief Title: Antiproteinuric Efficacy of Losartan Potassium in Patients With Non-Diabetic Proteinuric Renal Diseases (0954-213)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0954-213; MK0954-213; 2005_058
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Renal Disorder
MeSH Terms: conditions — Kidney Diseases | interventions — Losartan; Duration of Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0954, losartan potassium/Duration of Treatment: 20 weeks
Drug: Comparator: amlodipine / Duration of Treatment: 20 weeks

SUMMARY:
Antiproteinuric Efficacy of Losartan Potassium in Patients with Non-Diabetic Proteinuric Renal Diseases.

ELIGIBILITY:
Inclusion Criteria:

* Males or females at least 18 years of age with non-diabetic proteinuric renal diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2000-02; Primary Completion 2002-01 (Actual); Study Completion 2002-01 (Actual)

PRIMARY OUTCOMES:
24h proteinuria

SECONDARY OUTCOMES:
Changes in the plasma and urinary levels of TGF-beta

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Praga M, Andrade CF, Luno J, Arias M, Poveda R, Mora J, Prat MV, Rivera F, Galceran JM, Ara JM, Aguirre R, Bernis C, Marin R, Campistol JM. Antiproteinuric efficacy of losartan in comparison with amlodipine in non-diabetic proteinuric renal diseases: a double-blind, randomized clinical trial. Nephrol Dial Transplant. 2003 Sep;18(9):1806-13. doi: 10.1093/ndt/gfg284. PMID 12937228